#### PATIENT INFORMATION DOCUMENT:

**TITLE OF THE STUDY:** Multifactorial study of the relationship between the conditions of life and the incidence of risk of falling, from the Nursing perspective, in elderly adults of the Community.

Document date: 07/01/2018

PRINCIPAL RESEARCHER: Irene Escosura Alegre

#### **INTRODUCTION:**

You have been invited to participate in a research study. Please take the time you need to read the following information and consult what you need. Ask the researcher of this study if there is something that is not clear to you or if you want more information.

Aging involves a set of changes at the anatomical level and alterations in the systems, such as in the immune, neurological, endocrine, cardiovascular, digestive, respiratory, renal... Before these changes can occur the risk of dependence, fragility, disease... Appearing Geriatric Syndromes, including falls.

#### THE PURPOSE OF THE STUDY:

To study the relationship between living conditions and the incidence of risk of falls in older adults in the community.

### THE PROCESS:

An interview will take place during approximately half an hour. It will consist of asking you a series of questions that you should answer as faithfully as possible. You will also be weighed and measured.

Subsequently, we will go to the practical part, where five tests will be carried out: the Barthel Index (assessment of basic activities of daily life), the Downton fall risk assessment scale (for fall risk assessment), the Falls Efficacy Scale-International-FES-I- (to value the fear of falling), the Tinetti assessment tool (gait and balance assessment) and the Short Physical Performance Battery- SPPB- (for assessment of frailty and risk of disability and falls). They are short tests that do not require special skills to carry out.

In addition, medical and pharmacological records will be collected from your medical history.

## **ETHICAL AND LEGAL ASPECTS:**

Participation in this study would not cause any discomfort and does not imply any health risk.

All information obtained about you (questionnaires, surveys ...) will be coded under a unique number (the selection number) to guarantee anonymity. The code that identifies you will appear in each source of the study. Your identity will not be disclosed to any person. All information generated in this study will be used exclusively for the purposes specified here.

You can freely decide whether or not to participate in this study, participation is completely voluntary. If you decide to participate, you still have the possibility of withdrawing at any time and without having to give explanations, and without any penalty or negative consequences for you. Your decision to withdraw will not affect you at all. If you decide to participate, you must commit to doing the best possible as directed by the research team.

## **POSSIBLE BENEFITS:**

In case that you may can not directly benefit from your participation in this study, you will be collaborating in the development of scientific knowledge in the field of Health.

# **INFORMED CONSENT**

| TITLE OF THE STUDY Multifactorial study of the relationship between the conditions of life and the incidence of risk of falling, from the Nursing perspective, in elderly adults of the Community. |
|---|
| I (NAME AND SURNAME) |
| I have read the information document given to me. |
| I have been able to ask the questions about the study. |
| I have received enough information about the study. |
| I have spoken with (Name of the researcher) |
| I understand that participation is voluntary. |
| I understand that I can withdraw from the study: |
| a) When I want |
| b) Without having to give explanations |
| c) Without this having an impact on my rights and medical care. |
| I voluntarily agree to participate in the Project and authorize the use of all information obtained. I understand that I will receive a signed copy of this informed consent. |
| Date: |
| Signature of the participant |
| Signature of the researcher |